CLINICAL TRIAL: NCT06029790
Title: The Effect of Chewing Gum on Nausea, Vomiting and Bowel Functions After Colorectal Surgery: A Randomized Clinical Study
Brief Title: The Effect of Chewing Gum on Nausea, Vomiting and Bowel Function After Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Collaborators: Tarsus University (Other)
Responsible Party: Principal Investigator, Derya Gezer, Assistant Profesor, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CRC
Record Dates: First submitted 2023-08-28; First posted 2023-09-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Postsurgical Ileus
Keywords: postsurgical ileus; chewing gum; colorectal surgery
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, single-blind, parallel-group, randomized controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gum chewing (Experimental): All participants will receive standard postoperative care, 2 L/min of oxygen delivered via nasal cannula if oxygen saturation is below 95%. In addition, participants will be encouraged to use the incentive spirometer 10 times per hour to prevent respiratory complications such as pneumonia. In the postoperative period, all participants will be removed from bed and mobilized as soon as possible.
  For the patients in the experimental group, sugar-free xylitol gum containing 1.2-1.37 grams of xylitol per piece, available in the market, will be used. Participants in the experimental group will start chewing gum on the first postoperative day and will be allowed to chew a single piece of gum 3 times a day at 9:00, 14:00 and 19:00, respectively, for 15 minutes. The gum will be given to the participants regularly by a researcher until the first reported flatulence.
  Interventions: Other: gum chewing
- control group (No Intervention): All participants will receive standard postoperative care, 2 L/min of oxygen delivered via nasal cannula if oxygen saturation is below 95%. In addition, participants will be encouraged to use the incentive spirometer 10 times per hour to prevent respiratory complications such as pneumonia. In the postoperative period, all participants will be removed from bed and mobilized as soon as possible.
  The control group will receive only standard care.

INTERVENTIONS:
Other: gum chewing — For the patients in the experimental group, sugar-free xylitol gum containing 1.2-1.37 grams of xylitol per piece, available in the market, will be used. Participants in the experimental group will start chewing gum on the first postoperative day and will be allowed to chew a single piece of gum 3 times a day at 9:00, 14:00 and 19:00, respectively, for 15 minutes. The gum will be given to the participants regularly by a researcher until the first reported flatulence.
  Arms: gum chewing

SUMMARY:
False feeding refers to promoting gastrointestinal peristalsis by seeing, smelling, chewing, and tasting food, not getting food into the gastrointestinal tract. Postoperative sham feeding uses gum to promote the healing of gastrointestinal peristalsis. Although not fully understood, the physiological theory underlying gum chewing (fake feeding) to stimulate peristalsis and reduce postoperative intestinal recovery time is that the oral and chewing stimulation provided by chewing gum stimulates a neurohumoral reflex that increases gastrointestinal fluid secretion. This increases gastrointestinal motility. In addition, oral stimulation and chewing can stimulate the vagus nerve, which is also involved in promoting peristalsis. Finally, none of the existing theories adequately explain the effect of chewing/gum chewing on reducing postoperative inflammation in the gut, which may result in a reduced incidence of postoperative infection. In previous studies, physiological changes associated with gum appear to promote normal gastrointestinal function and subsequent postoperative/anesthetic recovery. Although many studies have been conducted to examine the effectiveness of chewing gum in patients undergoing colorectal resection, the results have been inconsistent. This can be attributed to differences in intestinal injuries affecting bowel function, differences in time under anesthesia and differences in anesthetics or pain control agents used for pain control affecting bowel function, and recovery time of peristalsis. Given the many factors known to affect postoperative ileus, chewing gum as an intervention remains a safe, accessible, and inexpensive option that remains to be explored.

DETAILED DESCRIPTION:
False feeding refers to promoting gastrointestinal peristalsis by seeing, smelling, chewing and tasting food, not getting food into the gastrointestinal tract. Postoperative sham feeding uses gum to promote healing of gastrointestinal peristalsis. Although not fully understood, the physiological theory underlying gum chewing (fake feeding) to stimulate peristalsis and reduce postoperative intestinal recovery time is that the oral and chewing stimulation provided by chewing gum stimulates a neurohumoral reflex that increases gastrointestinal fluid secretion. This increases gastrointestinal motility. In addition, oral stimulation and chewing can stimulate the vagus nerve, which is also involved in promoting peristalsis. Finally, none of the existing theories adequately explain the effect of chewing/gum chewing on reducing postoperative inflammation in the gut, which may result in a reduced incidence of postoperative infection. Previous studies have shown that physiological changes associated with gum support normal gastrointestinal function and subsequent postoperative/anesthetic recovery.

Some studies have shown that chewing gum after colorectal resection reduces postoperative flatulence and defecation time. showed that it reduces the risk of postoperative ileus. In contrast, some studies in patients undergoing open abdominal surgery or laparoscopy for various types of colorectal resection have shown no effect of chewing gum on postoperative first flatulence and time to defecation, has no significant effect in reducing the average hospital stay and has no significant effect in preventing postoperative nausea, vomiting, or bloating.

One possible reason for the inconsistent results of sham feeding using chewing gum to reduce the incidence of postoperative ileus may be differences in underlying colorectal cancer types and heterogeneity between surgical and postoperative care methods.

Although many studies have been conducted to examine the effectiveness of chewing gum in patients undergoing colorectal resection, the results have been inconsistent. This can be attributed to differences in intestinal injuries affecting bowel function, differences in time under anesthesia differences in anesthetics or pain control agents used for pain control affecting bowel function, and recovery time of peristalsis. Given the many factors known to affect postoperative ileus, chewing gum as an intervention remains a safe, accessible, and inexpensive option that remains to be explored. This study will provide empirical evidence that contributes to a body of literature supporting gum administration for affecting postoperative nausea, flatulence, and stool output in a well-defined sample.

Many interventions and strategies have been used to manage postoperative ileus, such as prokinetic agents and epidural anesthesia. However, these methods have limited efficacy and still have a relatively high incidence of postoperative ileus. Alternatively, chewing gum promotes gastrointestinal peristalsis in post-surgery patients without the adverse effects associated with early feeding. However, results in studies investigating the effect of chewing gum on postoperative recovery of gastrointestinal function after colorectal surgery are conflicting.

ELIGIBILITY:
Inclusion Criteria: Being over 18 years old,

* To have applied for elective colorectal surgery,
* Having undergone laparoscopic colorectal surgery,
* Not having a nasogastric insertion,
* Not having a vision-hearing problem,
* ECOG performance score to be between 0-2,

Exclusion Criteria:

* Performing emergency surgical intervention,
* Open colorectal surgery
* Need for intensive care after surgery,
* Stoma has been opened

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
prevention of postoperative ileus | 72 hours
  The first postoperative gas removal time and the first postoperative stool removal time will be questioned by the researcher. There is no standard scale for this.
Prevention of nausea-vomiting. | 72 saat
  Nausea and Vomiting Evaluation Form. In our study, PONV status will be evaluated as "Yes/No" at 0, 2, 4, 8, 12 and 24 hours using the Nausea and Vomiting Evaluation Form.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Results on the effects of chewing gum on nausea, vomiting and bowel functions after colorectal surgery will be shared. However, personal information will not be shared.

REFERENCES:
- [Background] van den Heijkant TC, Costes LM, van der Lee DG, Aerts B, Osinga-de Jong M, Rutten HR, Hulsewe KW, de Jonge WJ, Buurman WA, Luyer MD. Randomized clinical trial of the effect of gum chewing on postoperative ileus and inflammation in colorectal surgery. Br J Surg. 2015 Feb;102(3):202-11. doi: 10.1002/bjs.9691. Epub 2014 Dec 18. PMID 25524125
- [Background] Yang P, Long WJ, Wei L. Chewing Xylitol Gum could Accelerate Bowel motility Recovery after Elective Open Proctectomy for Rectal Cancer. Rev Invest Clin. 2018;70(1):53-58. doi: 10.24875/RIC.18002428. PMID 29513303
- [Background] Liu Q, Jiang H, Xu D, Jin J. Effect of gum chewing on ameliorating ileus following colorectal surgery: A meta-analysis of 18 randomized controlled trials. Int J Surg. 2017 Nov;47:107-115. doi: 10.1016/j.ijsu.2017.07.107. Epub 2017 Sep 1. PMID 28867465
- [Background] Hsu YC, Szu SY. Effects of Gum Chewing on Recovery From Postoperative Ileus: A Randomized Clinical Trail. J Nurs Res. 2022 Oct 1;30(5):e233. doi: 10.1097/jnr.0000000000000510. PMID 35951432
- [Background] Lee JT, Hsieh MH, Cheng PJ, Lin JR. The Role of Xylitol Gum Chewing in Restoring Postoperative Bowel Activity After Cesarean Section. Biol Res Nurs. 2016 Mar;18(2):167-72. doi: 10.1177/1099800415592966. Epub 2015 Jul 7. PMID 26156002
- [Background] Forrester DA, Doyle-Munoz J, McTigue T, D'Andrea S, Natale-Ryan A. The efficacy of gum chewing in reducing postoperative ileus: a multisite randomized controlled trial. J Wound Ostomy Continence Nurs. 2014 May-Jun;41(3):227-32. doi: 10.1097/WON.0000000000000019. PMID 24621587
- [Background] Kobayashi T, Masaki T, Kogawa K, Matsuoka H, Sugiyama M. Efficacy of Gum Chewing on Bowel Movement After Open Colectomy for Left-Sided Colorectal Cancer: A Randomized Clinical Trial. Dis Colon Rectum. 2015 Nov;58(11):1058-63. doi: 10.1097/DCR.0000000000000452. PMID 26445178
- [Background] Suh SY, Leblanc TW, Shelby RA, Samsa GP, Abernethy AP. Longitudinal patient-reported performance status assessment in the cancer clinic is feasible and prognostic. J Oncol Pract. 2011 Nov;7(6):374-81. doi: 10.1200/JOP.2011.000434. PMID 22379420
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Derived] Gezer D, Alptekin D, Yalav O, Eray IC. Effect of gum chewing on the return of bowel sounds, time to first flatus, and defecation after colorectal cancer surgery: A prospective, randomized controlled trial. Eur J Oncol Nurs. 2025 Dec;79:103039. doi: 10.1016/j.ejon.2025.103039. Epub 2025 Nov 7. PMID 41232231
- See also: Chewing gum for postoperative ileus after colorectal surgery: A systematic review of overlapping meta-analyses — https://doi.org/10.1016/j.cnre.2017.02.001